## **Cover Page**

## Participant Consent Form

Study Title: Unilateral Strength Training and Mirror Therapy for Enhancing Upper Limb Motor

Function Post Stroke: A Pilot Randomised Controlled Trial

Document creation date: March 20<sup>th</sup> 2015

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]

## **Participation Consent Form**

## Unilateral Strength Training and Mirror Therapy for Enhancing Upper Limb Motor Function Post Stroke: A Pilot Randomised Controlled Trial

| 1. | I confirm that I have received a copy of the Information Sheet for the above study. I have read it and I understand it. I have received an explanation of the nature and purpose of the study and what my involvement will be. | | |
|---|---|---|---|
| 2. | . I have had time to consider whet to ask questions. | her to take part in this study ar | nd I have had the opportunity |
| 3. | . I understand that my participatio research at any time. | n is voluntary and that I can de | cide to opt out of the |
| 4. | I understand that all information gathered about me during this study will be treated with full confidentiality. | | |
| 5. | I agree to the video recording of training sessions and understand that all recordings will be kept confidential. | | |
| 6. | . I agree to take part in the above : | study. | |
| Name of patient | | Date | Signature |